

# **Informed Consent**

English Title of the Study: Investigation of Possible Effects of a Lifestyle Product in a Double-blind Pre- Post-Between-Groups Study

German Title of the Study: Untersuchung möglicher Effekte eines Lifestyle-Produktes und Zusammenhänge von Persönlichkeits- und Intelligenzfaktoren mit paranormalen Überzeugungen in einer doppel-blinden Pre-Post-Between-Groups Studie

NCT number not available

Date 20.09.2020, Stuttgart

Principal Investigator Katharina Lingelbach, MSc

University of Stuttgart and Fraunhofer IAO

Stuttgart, Germany

ClinicalTrials.gov Protocol ID WAVEGUARD STRESS HUMANS FR01

Author Katharina Lingelbach, MSc

Version Draft 0.0



# Informed Consent of the study "Investigation of the stability of psychological states" - Time 1

Contact person:

Katharina, Lingelbach, M.Sc. mobile: +49 711 970-5342 katharina.lingelbach@iao.fraunhofer.de

### Dear participants,

Hereby, we would like to give you basic information about the procedure as well as the expected benefits and possible risks of the examination. If you have any difficulties in understanding the information, you can always ask the investigator-in-charge\*.

## Aim and benefits of the study

In this study we investigate psychological states over a period of one week.

For this purpose we will measure the activity of your brain, heart and the skin conduction resistance on your skin during a state of rest (relaxation). Afterwards we will ask you to fill in some questionnaires about your state of health and your personality.

The study is part of an industrial project to investigate a product as contract research. Unfortunately, we cannot give you some information at this time, as this knowledge could influence the results of the study. We will inform you about all risks in advance and you will be informed in detail at the end of the study, i.e. at the end of the second appointment.

# Procedure of the study

A total of 90 subjects will participate in the study. Participants will be randomly assigned to three different groups, with two groups participating in one intervention and one group corresponding to a control group for the collection of normative values. The assignment to the groups is double-blind, which means that neither the investigators\*in nor you know to which groups you will belong.

## Information on the current procedure

| 1 Study information + informed consent | 10 min |
|---|---|
| 2 questionnaires on sleep quality and current fatigue | 10 min |
| 3 Preparation of rest measurement | 30 min |
| 4 Resting measurement of brain and heart activity and skin conductance | 20 min |
| 5 Break | 10 min |
| 6 personality questionnaires | 10 min |
| 7 Conclusive thinking test | 30 min |
| 8 Break | 10 min |

9 Scale on paranormal beliefs and experiences, questionnaire on openness to complementary and alternative medicine, questionnaires on well-being, life satisfaction, positive and negative emotional states, anxiety and depression, stress perception and resilience 50 min



If you are interested in the study and agree to participate after detailed information about its procedure and conditions, the electrodes of the electroencephalography (EEG) will be attached to an EEG cap with the help of an electrode gel. With the help of these brain signals we are able to analyze the bioelectrical signals of the brain. Furthermore, measurements of physiological excitation are obtained by means of electrodermal activity and electrocardiography. The sensors for the measurement are attached to your finger and by means of a chest strap to your upper body.

The neurophysiological signals will be measured only during the 15 minutes of rest, after which we will remove the electrodes. All these examinations are risk-free and painless. All medical devices used in the study are CE-certified and have been extensively tested for safety.

After today's appointment, you will be asked to fill in some questions about your daily condition for the next 7 days. You can fill out the questions on your computer using your own ID and an online link. Your ID consists of a key of the

2nd and 3rd letter of the mother's first name / month of birth / 1st and 2nd letter of the street name

Example: Marta Mustermann / 01.01.1990 / Musterstraße 1 ID: ar01mu

If you have any questions during the 7 days, employees of the Universität Stuttgart and Fraunhofer IAO will support you via WhatsApp and email.

After the 7 days you will be invited back to the institute for a second appointment. For the second appointment you will again be informed about the study and your rights. If you attend the second appointment, you will receive another 50 € compensation. We will inform you again at your second appointment and ask you to sign the consent form again.

### Voluntary participation and withdrawal

This study will be conducted in accordance with current scientific and ethical guidelines. Your participation in this study is voluntary. If you choose not to participate in this study, you will not suffer any disadvantages. The same applies if you withdraw your consent at a later date. You have this option at any time. You do not have to give reasons for withdrawing your consent or withdrawing from the study.

## Risks

No external current is used to conduct the brain waves. The EEG, EDA, and ECG are non-invasive and stress-free measurements which are widely used worldwide, with no side effects and no safety risks to be expected. The examination is therefore completely safe for you. No invasive methods are used, i.e. we do not take blood or tissue samples. The data is used exclusively for research purposes.

### **Data protection**

All collected data is stored on magneto-optical disks. The recorded personal data is then pseudonymized (in the form of a multi-digit identification number) and stored without personal identification. During further processing and analysis of the data, only the identification number is used, so that the assignment between data and individual test persons cannot take place and misuse is impossible. The data is used exclusively for research purposes. Questionnaire and other analog data are digitized. The analog raw data are kept in a lockable cabinet, all digital data are stored centrally on a password-protected computer in the same room to which only the project managers mentioned below have access. The scientific evaluation of the pseudonymized data is initially carried out by Fraunhofer IAO. Further, the data will be scientifically evaluated by employees of the Universities of Stuttgart and Vienna. In the second case, the data is made available without any personal reference being established by the recipients. The data processing is carried out on the legal basis of Art. 6 para. 1 DSGVO. Your personal data will not be disclosed to third parties, third countries or international organizations. After the end of the project, the personal data (the name, address and account details for remuneration) will be stored exclusively in accordance with Art. 6 para. 1 sentence 1 lit. c) DSGVO in accordance with the storage regulations of the relevant tax legislation and will be deleted after 10 years as soon as legally permissible. The personal data will be blocked for deviating processing after the end of the project and the re-identification list, which



allows the assignment of the personal reference to the pseudonymized study data used for research, will be destroyed at the earliest possible time after the end of the project. The previously personal study data are irreversibly made fully anonymous from this point on. The fully anonymized data will be further processed and analyzed by scientific staff of the University of Stuttgart, Vienna and Fraunhofer IAO. Until full anonymization has taken place, the final deletion of your own data can be requested from Fraunhofer IAO at any time. The deletion of data from both sessions (Session 1 and Session 2) or one session each (Session 1 or Session 2) can be requested.

The legal basis for the processing of personal data in clinical studies or studies on humans is your written consent in accordance with the German Data Protection Act (DSGVO), the Declaration of Helsinki (Declaration of the World Medical Association on the Ethical Principles of Medical Research on Humans) and the Guideline for Good Clinical Practice. For clinical trials with medicinal products, the German Medicines Act and for clinical trials with medical devices, the Medical Devices Act must also be applied. At the same time as the DSGVO, the revised Federal Data Protection Act (BDSG-neu) and state data protection regulations come into force in Germany.

You have the following rights regarding your data:

# Consent to the processing of personal data and right of revocation

The processing of your personal data is only lawful with your consent. You have the right to revoke your consent to the processing of personal data at any time without giving reasons. However, the data collected up to this point may be processed by the authorities named in the subject information or declaration of consent for the respective study. If you revoke your consent, the lawfulness of the processing carried out on the basis of your consent until revocation remains unaffected.

### Right to information, correction, deletion, etc.

You are entitled to so-called data subject rights, i.e. rights that you can exercise as a data subject in individual cases. You can assert these rights against the University of Würzburg. They result from the DSGVO.

### Right to information, Art. 15 DSGVO

You have the right to be informed about your personal data that has been collected, processed or, if applicable, transferred to third parties in the course of the study.

# Right of rectification, Art. 16 DSGVO

If you discover that incorrect data concerning your person is being processed, you can request a correction. Incomplete data must be completed taking into account the purpose of the processing.

### Right of cancellation, Art 17 DSGVO

You have the right to have your personal data deleted if there are certain reasons for deletion. This is particularly the case if they are no longer necessary for the purpose for which they were originally collected or processed or if you revoke your consent.

### Right to limitation of processing, Art. 18 DSGVO

You have the right to limit the processing of your data. This means that your data will not be deleted, but will be marked in order to limit its further processing or use.

# Right to data transferability, Art. 20 DSGVO

You have the right to request the personal data concerning you that you have provided to us in a standard electronic format.



They have a general right of objection even against legitimate data processing that is in the public interest, in the exercise of official authority or on the basis of the legitimate interest of a body.

If you wish to exercise one of these rights, please contact the experimenter mentioned below. You also have the right to lodge a complaint with the data protection supervisory authority(ies) if you believe that the processing of personal data concerning you is in breach of the DSGVO. You may lodge a complaint with the supervisory authority informally with the Fraunhofer data protection officer (email: datenschutz@zv.fraunhofer.de).

### Further clarification after completion of the study

In this study, some information was withheld because it would affect the results of the study. However, they were informed about all risks of participation.

At the end of the study, i.e. after the end of the second appointment or if the study is terminated, you will receive a comprehensive explanation of the study contents.

Should you have any difficulties in understanding the study or have any questions, you can always ask the investigator. Thank you very much for your interest and cooperation!

# **Subject information - Time 1 Declaration of consent**

to participate in the study "Investigation of the stability of psychological states"

With this signature I confirm that I have been informed about the nature, significance and scope, personal advantages and disadvantages, risks, potential complications and side effects of the above-mentioned study. I am participating in the study voluntarily and have been informed that I can terminate my participation in the study at any time and without giving any further reasons and that I will not suffer any disadvantages as a result.

I have been informed about the handling of the personal data collected in the study and any additional questions have been answered to my satisfaction. The data will be stored in accordance with the applicable data protection regulations. Only Fraunhofer IAO staff\* involved in the project have access to the personal data. They are subject to the obligation of secrecy. The fully anonymized data will be processed and scientifically evaluated by scientific staff members of the Universities of Vienna and Stuttgart. Personal data will not be passed on to third parties.

| processing of personal data. |
|------------------------------------------------------|
| Place, date Signature of study participant |
| Place, date Signature of study/experimental director |

I hereby confirm my voluntary participation in the study and consent to the collection and



# Patient information on the handling of the product within the scope of the study "Investigation of the stability of psychological states"

Contact person:

Katharina, Lingelbach, M.Sc. mobile: +49 711 970-5342 katharina.lingelbach@iao.fraunhofer.de

After your first appointment at the Fraunhofer IAO you will receive the product to be examined in this study on loan at your home for the period of the study.

### Positioning of the product

For our study it is very important that you have the product in your area within the next 7 days. You should position it at a maximum distance of 2 meters from your body. Position the product in a safe and dry place. It is best to place the product during the day, on your desk and at night on your bedside table. It should stand upright and not be exposed to extreme temperatures or moisture. No other objects (such as the PC, cell phone, decorative items, cables, wifi router or alarm clock) should be placed within a radius of 25 cm and it should stand freely at a distance of 25 cm from the wall in the room. Please do not place anything on the product. This is very important for the results of our study.

### On the way

If you are on the road a lot or have to do business over several hours, you can take the product with you safely protected in a protective bag. It weighs about 850 g.

We ask you to handle the product with care and attention, as you should return it to us undamaged and in its original condition after the end of the study. If you have pets or children, please place the product out of reach.

### Handing over the product on termination or the second session

Please bring the product to your second appointment undamaged and in its original condition to return it to us. In case you forgot the product, we ask you to return it within the next 2 days. We will transfer the money to your account only after you have returned the product. If you wish to voluntarily stop the study, we ask you to return the product within the next two days.

### Risks

The product examined here is a TÜV-certified lifestyle product that does not emit electromagnetic radiation and has no invasive influence on your body. Furthermore, no toxic or electronic components (e.g. camera and microphones) are built into the product. When used properly, the product poses no health risks. Even if the product should be damaged, there are no particular risks. In case you notice any negative effects of the product, please inform us. We will provide you with the contact details of the manufacturer and you can contact them.

### Questionnaires

Every day we will ask you to fill in some questions about your daily condition. You can fill out the questions on your computer using your own ID and an online link. We will send you the online link either by email or by WhatsApp.

Your ID consists of a key of the 2nd and 3rd letter of the mother's first name / month of birth / 1st and 2nd letter of the street name.

Example: Marta Mustermann / 01.01.1990 / Musterstraße 1 ID: ar01mu

At this time, we are unfortunately unable to provide you with some information as this knowledge may influence the results of the study. We will inform you about all risks in advance and you will be informed



in detail after the end of the study, i.e. at the end of the second appointment. We assure you that the product is harmless and poses no risks if handled properly. For our study it is important that you carry the product with you for as long as possible and with a maximum distance of 2 meters.

If you have any questions during the 7 days, employees of the University of Stuttgart and Fraunhofer IAO will support you via WhatsApp and via email.

## Voluntary participation and resignation

This study will be conducted in accordance with current scientific and ethical guidelines. Your participation in this study is voluntary. If you choose not to participate in this study, you will not suffer any disadvantages. The same applies if you withdraw your consent at a later date. You have this option at any time during these 7 days and after the subsequent clarification of the study objectives. You do not have to give reasons for withdrawing your consent or withdrawing from the study.

Should you have any difficulties or questions, you can always ask the experimenter.

# Thank you for your interest and cooperation!

Subject information - Handling of the product

Declaration of consent

to participate in the study "Investigation of the stability of psychological states"

With this signature I confirm that I have been informed about the nature, significance and scope, personal advantages and disadvantages, risks, potential complications and side effects of the above-mentioned study. I am participating in the study voluntarily and have been informed that I can terminate my participation in the study at any time and without giving any further reasons and that I will not suffer any disadvantages as a result.

I also confirm that I have received the product under investigation here. I confirm that I have received the test person information and handling of the product and have read it carefully. I assure that I will return the product received undamaged at the second appointment.

I hereby confirm my voluntary participation in the study and consent to the collection and processing of personal data.

| Place, date Signature of study participant |
|------------------------------------------------------|
| Place, date Signature of study/experimental director |



# Informed Consent of the study "Investigation of the stability of psychological states" - Time 2

Contact person:

Katharina, Lingelbach, M.Sc. mobile: +49 711 970-5342 katharina.lingelbach@iao.fraunhofer.de

### Dear participants,

Welcome to our second trial date. With this information sheet we would like to give you again basic information about the procedure as well as the expected benefits and possible risks of the study. Should you have any difficulties in understanding the information, please do not hesitate to ask the investigator-in-charge.

### Aim and benefits of the study

In this study we investigate psychological states over a period of one week.

For this purpose, we will measure again today the activity of your brain, heart and the skin conduction resistance on your skin during a state of rest (relaxation). Afterwards we will ask you to fill in some questionnaires about your state of health and your personality, just like the first time.

The study is part of an industrial project to investigate a product as contract research. Unfortunately, we cannot give you any information at this time, as this knowledge could influence the results of the study. We will inform you about all risks in advance and you will be informed in detail at the end of the study, i.e. at the end of the second appointment.

## Procedure of the study

A total of 90 subjects will participate in the study. Participants will be randomly assigned to three different groups, with two groups participating in one intervention and one group corresponding to a control group for the collection of normative values. The assignment to the groups is double-blind, which means that neither the investigators\*in nor you know to which groups you will belong.

### Information on the current procedure

| 1 Study information + informed consent | 10 min |
|---|---|
| 2 questionnaires on well-being, stress and special events | 10 min |
| 3 questionnaires on sleep quality and current fatigue | 10 min |
| 4 Preparation of rest measurement | 30 min |
| 5 Resting measurement of brain and heart activity and skin conductance | 20 min |
| 6 Break | 10 min |
| 7 Scale on paranormal beliefs and experiences, questionnaire on openness to complementary and alternative medicine, questionnaires on well-being, life satisfaction, positive and negative emotional states, anyiety and depression, class, persention, and recilianse. | |
| states, anxiety and depression, stress perception and resilience | 50 min |
| 8 questionnaires on fear of radiation, electromagnetic hypersensitivity | 10 min |
| TI 11 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |

The appointment today usually takes about 3 hours. It is remunerated with 50 €.

If you are interested in the study and agree to participate after detailed information about its procedure and conditions, the electrodes of the electroencephalography (EEG) will be attached to an EEG cap with



the help of an electrode gel. With the help of these brain signals we are able to analyze the bioelectrical signals of the brain. Furthermore, measurements of physiological excitation are obtained by means of electrodermal activity and electrocardiography. The sensors for the measurement are attached to your finger and by means of a chest strap to your upper body.

The neurophysiological signals will be measured only during the 15 minutes of rest, after which we will remove the electrodes. All these examinations are risk-free and painless. All medical devices used in the study are CE-certified and have been extensively tested for safety.

## Voluntary participation and withdrawal

This study will be conducted in accordance with current scientific and ethical guidelines. Your participation in this study is voluntary. If you choose not to participate in this study, you will not suffer any disadvantages. The same applies if you withdraw your consent at a later date. You have this option at any time. You do not have to give reasons for withdrawing your consent or withdrawing from the study.

#### Risks

No external current is used to conduct the brain waves. The EEG, EDA, and ECG are non-invasive and stress-free measurements which are widely used worldwide, with no side effects and no safety risks to be expected. The examination is therefore completely safe for you. No invasive methods are used, i.e. we do not take blood or tissue samples. The data is used exclusively for research purposes.

### **Data protection**

All collected data is stored on magneto-optical disks. The recorded personal data is then pseudonymized (in the form of a multi-digit identification number) and stored without personal identification. During further processing and analysis of the data, only the identification number is used, so that the assignment between data and individual test persons cannot take place and misuse is impossible. The data is used exclusively for research purposes. Questionnaire and other analog data are digitized. The analog raw data are kept in a lockable cabinet, all digital data are stored centrally on a password-protected computer in the same room to which only the project managers mentioned below have access. The scientific evaluation of the pseudonymized data is initially carried out by Fraunhofer IAO. Further, the data will be scientifically evaluated by employees of the Universities of Stuttgart and Vienna. In the second case, the data is made available without any personal reference being established by the recipients. The data processing is carried out on the legal basis of Art. 6 para. 1 DSGVO. Your personal data will not be disclosed to third parties, third countries or international organizations. After the end of the project, the personal data (the name, address and account details for remuneration) will be stored exclusively in accordance with Art. 6 para. 1 sentence 1 lit. c) DSGVO in accordance with the storage regulations of the relevant tax legislation and will be deleted after 10 years as soon as legally permissible. The personal data will be blocked for deviating processing after the end of the project and the re-identification list, which allows the assignment of the personal reference to the pseudonymized study data used for research, will be destroyed at the earliest possible time after the end of the project. The previously personal study data are irreversibly made fully anonymous from this point on. The fully anonymized data will be further processed and analyzed by scientific staff of the University of Stuttgart, Vienna and Fraunhofer IAO. Until full anonymization has taken place, the final deletion of your own data can be requested from Fraunhofer IAO at any time. The deletion of data from both sessions (Session 1 and Session 2) or one session each (Session 1 or Session 2) can be requested.

The legal basis for the processing of personal data in clinical studies or studies on humans is your written consent in accordance with the German Data Protection Act (DSGVO), the Declaration of Helsinki (Declaration of the World Medical Association on the Ethical Principles of Medical Research on Humans) and the Guideline for Good Clinical Practice. For clinical trials with medicinal products, the German Medicines Act and for clinical trials with medical devices, the Medical Devices Act must also be applied. At the same time as the DSGVO, the revised Federal Data Protection Act (BDSG-neu) and state data protection regulations come into force in Germany.

You have the following rights regarding your data:



### Consent to the processing of personal data and right of revocation

The processing of your personal data is only lawful with your consent. You have the right to revoke your consent to the processing of personal data at any time without giving reasons. However, the data collected up to this point may be processed by the authorities named in the subject information or declaration of consent for the respective study. If you revoke your consent, the lawfulness of the processing carried out on the basis of your consent until revocation remains unaffected.

## Right to information, correction, deletion, etc.

You are entitled to so-called data subject rights, i.e. rights that you can exercise as a data subject in individual cases. You can assert these rights against the University of Würzburg. They result from the DSGVO.

## Right to information, Art. 15 DSGVO

You have the right to be informed about your personal data that has been collected, processed or, if applicable, transferred to third parties in the course of the study.

### Right of rectification, Art. 16 DSGVO

If you discover that incorrect data concerning your person is being processed, you can request a correction. Incomplete data must be completed taking into account the purpose of the processing.

# Right of cancellation, Art 17 DSGVO

You have the right to have your personal data deleted if there are certain reasons for deletion. This is particularly the case if they are no longer necessary for the purpose for which they were originally collected or processed or if you revoke your consent.

### Right to limitation of processing, Art. 18 DSGVO

You have the right to limit the processing of your data. This means that your data will not be deleted, but will be marked in order to limit its further processing or use.

### Right to data transferability, Art. 20 DSGVO

You have the right to request the personal data concerning you that you have provided to us in a standard electronic format.

### Right to object to unacceptable data processing, Art. 21 DSGVO

They have a general right of objection even against legitimate data processing that is in the public interest, in the exercise of official authority or on the basis of the legitimate interest of a body.

If you wish to exercise one of these rights, please contact the experimenter mentioned below. You also have the right to lodge a complaint with the data protection supervisory authority(ies) if you believe that the processing of personal data concerning you is in breach of the DSGVO. You may lodge a complaint with the supervisory authority informally with the Fraunhofer data protection officer (email: datenschutz@zv.fraunhofer.de).

## Further clarification after completion of the study

In this study, some information was withheld because it would affect the results of the study. However, they were informed about all risks of participation.

At the end of the study, i.e. after the end of the second appointment or if the study is terminated, you will receive a comprehensive explanation of the study contents.

Should you have any difficulties in understanding the study or have any questions, you can always ask the investigator. Thank you very much for your interest and cooperation!



# **Subject information - Time 2 Declaration of consent**

to participate in the study "Investigation of the stability of psychological states"

With this signature I confirm that I have been informed about the nature, significance and scope, personal advantages and disadvantages, risks, potential complications and side effects of the above-mentioned study. I am participating in the study voluntarily and have been informed that I can terminate my participation in the study at any time and without giving any further reasons and that I will not suffer any disadvantages as a result.

I have been informed about the handling of the personal data collected in the study and any additional questions have been answered to my satisfaction. The data will be stored in accordance with the applicable data protection regulations. Only Fraunhofer IAO staff\* involved in the project have access to the personal data. They are subject to the obligation of secrecy. The fully anonymized data will be processed and scientifically evaluated by scientific staff members of the Universities of Vienna and Stuttgart. Personal data will not be passed on to third parties.

I hereby confirm my voluntary participation in the study and consent to the collection and processing of personal data.

Place, date Signature of study participant Place, date Signature of study/experimental director



# Post-experimental debriefing of the study objectives

# Investigation of Possible Effects of a Lifestyle Product in a Doubleblind Pre- Post-Between-Groups Study

Thank you very much for your participation in our study!

With this study we investigate whether the product Qi-Shield of the company Waveguard GmbH has effects on a subjective and neurophysiological level on certain physical and psychological conditions such as stress, sleep quality and well-being. The product has been developed for private and business use, with the aim of restoring a naturally balanced living environment, according to the company. According to the company Waveguard GmbH, the product contains conductive liquids in specific geometric configurations designed to interact with high frequency and environmental electromagnetic fields.

The Qi-Shield product is a TÜV-approved lifestyle product that does not emit electromagnetic radiation and has no invasive effect on your body. Furthermore, no electronic components (e.g. camera and microphones) are built into the product. Further descriptions of the product can be found on the company's homepage: https://www.waveguard.com/startseite

We would like to emphasize here that we do not take any responsibility for the correctness of the statements on the website. Furthermore, the study does not serve as a recommendation of the products of Waveguard GmbH.

The industry partner assumes that the device has positive psychological and physical effects on humans after a certain exposure time of 7 days.

We have investigated this statement by means of an "between-group" study design with a pre-post-examination. There were three groups: a) group A received the Qi-Shield product with conductive fluids in geometric configuration, b) group B received the Qi-Shield product without conductive fluids in geometric configuration (this corresponds to a placebo group), and c) the last group did not receive any product in order to assess the pure effect of a test as a comparison.

In order to investigate a possible effect, we examine the comparability of the groups in different areas such as demographic data, statements on current well-being or even personality and attitudes towards paranormal beliefs and critical thinking. For a statistical comparison, the difference between the first and second measurement is calculated and compared between the different groups. If the product is effective, there should be a significant (significant) difference between group A and B with increased well-being, improved sleep quality and reduced stress perception.

In a further question we investigate possible connections between personality and intelligence factors with a tendency to paranormal beliefs. In the case of a placebo effect (i.e. that there is no significant difference between the two conditions A and B) we are interested in predicting the expression of the placebo effect using the personality and intelligence factors.

After the end of the project, the personal data (name, address and account details for remuneration) will be stored exclusively in accordance with Art. 6 para. 1 sentence 1 lit. c) DSGVO in accordance with the storage regulations of the relevant tax legislation and will be deleted after 10 years as soon as legally permissible. The personal data will be blocked for deviating processing after the end of the project and the re-identification list, which allows the assignment of the personal reference to the pseudonymized study data used for research, will be destroyed at the earliest possible time after the end of the project. The previously personal study data are irreversibly made fully anonymous from this point on. The fully anonymized data will be further processed and analyzed by scientific staff of the University of Stuttgart, Vienna and Fraunhofer IAO. If you request earlier deletion of the personal data, please contact the study director.



You will receive the amount of 100€ for your participation by bank transfer within the next 6 weeks.

### Voluntary participation and withdrawal

This study was conducted in compliance with the applicable scientific and ethical guidelines. Your participation in this study is voluntary. If you choose not to participate in this study, you will not suffer any disadvantages. This also applies if you revoke your consent after completion of the study or at a later date. You have this option at any time. You do not have to give reasons for withdrawing your consent or withdrawing from the study.

If you still have questions or if questions have arisen in the course of the study, you are welcome to contact the study director even after the study has ended.

Thank you for your interest and cooperation!

Study director and contact person:

Katharina, Lingelbach, M.Sc. Phone: +49 711 970-5342

katharina.lingelbach@iao.fraunhofer.de

As a general address at the institute, you can alternatively always use our email address proband-hci@iao.fraunhofer.de.

# Post-experimental debriefing Declaration of consent

to participate in the study "Investigation of the stability of psychological states" in the context of possible effects of the product Qi-Shield of the company Waveguard GmbH and to store and process the collected data.

With this signature I confirm that I have been informed about the nature, significance and scope, personal advantages and disadvantages, risks, potential complications and side effects of the above-mentioned study. I am participating in the study voluntarily and have been informed that I can terminate my participation in the study at any time and without giving any further reasons and that I will not suffer any disadvantages as a result.

I have been informed about the handling of the personal data collected in the study and any additional questions have been answered to my satisfaction. The data will be stored in accordance with the applicable data protection regulations. Only Fraunhofer IAO staff\* involved in the project have access to the personal data. They are subject to the obligation of secrecy. The fully anonymized data will be processed and scientifically evaluated by scientific staff members of the Universities of Vienna and Stuttgart. Personal data will not be passed on to third parties.

I hereby confirm my voluntary participation in the study and consent to the storage and processing of personal data.